CLINICAL TRIAL: NCT02958501
Title: Optimal Substitution Dose of the Vitamin D During Winter Time in Patient With Inflammatory Bowel Diseases (IBD)
Brief Title: Vitamin D Substitution During Winter Time
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Collaborators: Nemocnice T.Bati, Zlin (Unknown); Brno University Hospital (Other)
Responsible Party: Principal Investigator, MUDr. Jan Matous, Jan Matous, MD, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DV1607
Record Dates: First submitted 2016-11-01; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Vitamin D Substitution
Keywords: Vitamin D; Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IU/Day (Active Comparator): This is standard dose of the drug (colecalciferol), which is not calculated in relation to patient body weight
  Interventions: Drug: Colecalciferol
- IU/Kg/Day (Active Comparator): This is dose of the drug (colecalciferol), which is based or calculated in relation to patient actual body weight
  Interventions: Drug: Colecalciferol

INTERVENTIONS:
Drug: Colecalciferol — Drug

SUMMARY:
The purpose of this study is to confirm anticipated substitution dose of the vitamin D for sustained blood level during winter time in patients with inflammatory bowel diseases (IBD)

DETAILED DESCRIPTION:
Vitamin D substitution is widely recommended. Suggested substitution doses are increasing over the time. No exact body requirement is known for patients with IBD at present. Aim of the study was to confirm substitution dose obtained from model.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with inflammatory bowel disease

Exclusion Criteria:

* Liver disease
* Renal disease
* Hypercalcemia
* Hyperparathyreoidism
* Chronic pancreatitis
* Concomitant vitamin D medication
* Pregnancy
* Sarcoidosis
* Malignancy
* Inability to obtain valid data from subject

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in vitamin D blood level after follow-up interval | 4 Months
  Change of the D vitamin level after follow-up interval in groups substituted according to weight or in fixed daily dose.

SECONDARY OUTCOMES:
Change in vitamin D after follow-up interval according to weight | 4 Months
  Change in vitamin D after follow-up interval according to weight. Superiority of weight base dosing to fixed daily dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No